CLINICAL TRIAL: NCT00314730
Title: Outcomes in the Palm of Your Hand: Improving the Quality and Continuity of Patient Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government); Canadian Health Services Research Foundation (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 16402
Record Dates: First submitted 2006-04-13; First posted 2006-04-14 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Computers, Handheld; Outcomes Assessment, Patient

INTERVENTIONS:
Device: handheld Personal Digital Assistant (PDA)

SUMMARY:
This study evaluates the usability of personal digital assistants (PDAs) by nurses for collecting, utilizing and communicating patient health information, and the feasibility of using PDAs to increase nurses' access to and utilization of best-practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Nurses are eligible to participate if they work on a participating unit, 20 or more hours/week
* Patients are eligible if they are being cared for on a participating unit, are able to provide informed consent in English, and are able to answer questions about their daily activities and symptoms (pain, nausea, dyspnea, fatigue.)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2006-05; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
nursing communication and coordination
patient functional status
patient symptoms (pain, nausea, dyspnea, fatigue)
patient therapeutic self care

CONTACTS AND LOCATIONS:
Overall Officials: Diane Doran, PhD, RN, Principal Investigator — Professor, Faculty of Nursing, Univ of Toronto
Locations (3):
- Canada (3):
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - St. Joseph's Health Center, Toronto, Ontario